CLINICAL TRIAL: NCT00207909
Title: The Role of Hemodynamics, Cytokine Response, and Modulators of Apoptosis on Urine Output in Patients With Acute Renal Failure on CVVH
Brief Title: Study of Patients With Acute Renal Failure on CVVH
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 04-114; 06585
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Renal Failure
Keywords: Acute Renal Failure; Contiuous Veno Venous Hemofiltration
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Acute kidney failure is common in children in the Pediatric Intensive Care Unit (PICU). You are being asked to participate in this study because your child is being treated for kidney failure with continuous veno-venous hemofiltration (CVVH). CVVH is a continuous, gentle form of removing excess fluids and small wastes from the blood, similar to kidney dialysis (artificial kidney). It is an accepted therapy for temporary support of kidney failure. In some patients with acute kidney failure, beginning CVVH is followed by a temporary decrease of urine output. The reason why this happens is currently unknown. The purpose of this study is to determine why this happens.

DETAILED DESCRIPTION:
Acute renal failure is common in children in the pediatric intensive care unit. Renal replacement therapies such as peritoneal dialysis (PD), intermittent hemodialysis (IHD), and continuous venovenous hemofiltration (CVVH) have been used in the management of acute renal failure. CVVH is becoming increasingly utilized in pediatric acute renal failure. However, in patients who have acute renal failure, the institution of CVVH is often followed by a progression to oliguria or anuria. The underlying pathophysiology of this change is unknown. We believe that this progression is influenced by changes in the renin-angiotensin axis, cytokine response, and other modifiers of renal hemodynamics. By serially measuring components of those systems, this study will attempt to elucidate the pathophysiology of the decreased urine output seen with institution of CVVH. Once this process is understood, future studies should focus on prevention and treatment of this complication.

General Hypothesis

The decrease in urine output seen after the initiation of CVVH is associated with increased angiotensin converting enzyme (ACE) levels, increased renin activity, increased angiotensin II levels, increased atrial naturetic peptide (ANP) levels, increased endothelin-1 levels, increased arginine vasopressin (AVP) levels, and alterations of cytokine levels and modulators of apoptosis.

ELIGIBILITY:
Inclusion Criteria:

The general goal of patient selection is to enroll all children for whom CVVH is instituted.

Inclusion criteria:

Age

* 6 months -18 years old
* Patients less than 6 months of age on ECMO (addendum #1)

Indication for CVVH: including, but not limited to :

* Acute Renal Failure
* Oliguria
* Anuria
* Hyperkalemia
* Severe acidemia
* Azotemia
* Pulmonary Edema
* Uremic complications
* Severe electrolyte abnormalities
* Drug overdose with a filterable toxin
* Anasarca
* Rhabdomyolysis

Exclusion Criteria:

* Age

  * Less than 6 months old (unless on ECMO)
  * Greater than 18 years old Weight
  * Less than 5 kilograms (unless ON ECMO) Location
  * Cardiac Intensive Care Unit
  * Neonatal Intensive Care Unit

Non-adherence:

Inability or unwillingness of the legal guardian to provide consent or inability or unwillingness of the child to provide assent

Min Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients Pediatric Intensive Care Unit @ Egleston meeting inclusion criteria / avoiding exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2005-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine the underlying etiology of the decrease in urine output seen with the institution of CVVH by examining patient's physiologic hormonal responses. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James D Fortenberry, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States